CLINICAL TRIAL: NCT04537260
Title: How Will an Educational Video About the Induction of Labor Process Impact Patient's Knowledge of and Satisfaction With the Induction Process
Brief Title: An Educational Video's Impact on the Induction of Labor Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NCR191281
Record Dates: First submitted 2020-08-25; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Knowledge; Satisfaction, Patient
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Participants were either enrolled in the control arm (no intervention) or the intervention group (3-minute educational video intervention)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The research member enrolling the patient in the study, the participant, and the person collecting the questionnaires were all blind to what arm of the study the participant would be placed into (control vs intervention with video group). A computer-generated allocation sequence to determine randomization. Randomization assignments were placed in sealed, opaque envelopes that were opened sequentially after verbal and signed consent was obtained for the study. The research team members who collected the outcome data (example, parity, delivery method, etc) was also blind to which arm the participant was assigned too.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Standard of Care) (No Intervention): The control group took the knowledge-based survey about induction of labor prior to meeting their provider (midwife or obstetrician) on the day of scheduled induction. Twenty-four to forty-eight hours after delivery, at a time convenient to the participant during the postpartum stay at GW, a research team member asked the participant to fill out a second survey, focused on satisfaction with the labor and delivery process.
- Intervention Arm (Educational video) (Experimental): The intervention group had the opportunity to watch the 3-minute educational video. The video shown to these participants is linked here: https://youtu.be/Pc9tcIV4Dm8. After watching the video, the participant was asked to take the knowledge-based survey. Twenty-four to forty-eight hours after delivery, at a time convenient to the participant during the postpartum stay at GW, a research team member asked the participant to fill out a second survey, focused on satisfaction.
  Interventions: Behavioral: Educational Video

INTERVENTIONS:
Behavioral: Educational Video — Those in the intervention arm were asked to watch the 3-minute educational video prior to the knowledge questionnaire and meeting their provider (midwife or obstetrician). The video shown to these participants is linked here: https://youtu.be/Pc9tcIV4Dm8.
  Arms: Intervention Arm (Educational video)

SUMMARY:
The investigators have created a brief, 3-minute video that discusses the induction of labor process. The aim of this study is to evaluate, via a randomized method, how this educational video impact's patients' knowledge and satisfaction with the induction of labor process.

Purpose: Evaluate how an educational video impacts patients' knowledge and satisfaction with the induction of labor process

Research questions:

1. Does a brief educational video improve patients' baseline knowledge of the induction of labor process when compared to patients' who receive traditional care?
2. Does a brief educational video improve patients' overall satisfaction with their delivery course when compared to patients' who received the standard care? Hypothesis: Those patients' shown a brief educational video will have a higher baseline knowledge about the induction process and higher satisfaction with their delivery course compared to patients who received the standard in-office counseling.

DETAILED DESCRIPTION:
Recruitment and Data Collection:

Patients were screened for study enrollment during routine prenatal visits at the George Washington University Hospital. A trained research team member met with and spoke to eligible patients about the randomized study at the time of their scheduled induction of labor visit. There was an induction of labor schedule that is created monthly, which the research team members had access to and determined when eligible participants had their induction of labor visit scheduled.

Informed consent was obtained from the patient if they were interested in participating. Privacy and confidentiality were assured as approved team members were the only individuals with access to patient records and maintained strict confidentiality. All consent forms were kept in a locked cabinet and survey responses were de-identified. Patients were able to ask questions and/or opt out of the study at any time.

The research team member assessed patient's understanding of the information and participation by asking them to describe in their own words what they were consenting to. Signed informed consent were obtained prior to study enrollment.

Once a patient was enrolled, they were randomized to the control group (no intervention) or the intervention group (3-minute educational video intervention). The randomization schedule was predetermined. The enrolled participant was given a pre-randomized study envelope that contained a unique Study ID number, randomization group, and paper surveys.

The control group took the knowledge-based survey. Twenty-four to forty-eight hours after delivery, at a time convenient to the participant during the postpartum stay at GW, a research team member asked the participant to fill out a second survey, focused on satisfaction with the labor and delivery process.

The intervention group had the opportunity to watch the 3-minute educational video. The video shown to these participants is linked here: https://youtu.be/Pc9tcIV4Dm8. After watching the video, the participant was asked to take the knowledge-based survey. Twenty-four to forty-eight hours after delivery, at a time convenient to the participant during the postpartum stay at GW, a research team member asked the participant to fill out a second survey, focused on satisfaction.

If the patient ultimately chose not to participate in the study following the signing of informed consent, all their data was destroyed. All of the surveys were stored in a locked cabinet, secured. No one but the research team members had access to the collected data and none of the stored paper copies had any identifying information. The basic demographic information, as well as the outcome of the induction of labor process, was collected using the hospital's electronic medical record. Some of the information (race and ethnicity) was collected by self-report. Emails were obtained by self-report on a voluntary basis. They were only collected if patients wished to be entered into the raffle for the Amazon gift card.

Recruitment goal:

At minimum, the goal was an n= of 106 total, 53 per arm. This was powered based on an alpha of 0.05, 80% power, 10% attrition rate to accurately detect a 20% difference given 96% correct in the intervention group.

Data entry:

After enrollment and completion of study surveys, a member of the research team entered in all of the information collected into a de-identified Redcap database using the unique Study ID numbers. The research team also collected data from the patient's electronic medical record about the enrolled participant's induction of labor process, including gravity, parity, pregnancy complications, induction agents utilized, and delivery method (vaginal vs cesarean delivery). All of this data was entered into the de-identified Redcap database. Access to the participant's medical record was only available to the research team through the MFA's HIPAA compliant, password protected, firewalled electronic medical record (Allscripts) and GW hospitals' EMR (Cerner).

After the data was entered into Redcap, a second and different member of the research team re-checked the entry to ensure the answers were correctly captured into the system.

Statistical Analysis:

The investigators used specific methods to address our hypothesis: Those patients' shown a brief educational video will have a higher baseline knowledge about the induction process and higher satisfaction with their delivery course compared to patients who received the standard in-office counseling.

1. Does a brief educational video improve patients' baseline knowledge of the induction of labor process when compared to patients' who receive the traditional care?

   The investigators used mean, standard deviation, and analysis via Mann-Whitney U tests.
2. Does a brief educational video improve patients' overall satisfaction with their delivery course when compared to patients' who received the standard care?

The investigators used mean, standard deviation, and analysis via Mann-Whitney U, Chi-Square, and Fisher's exact tests.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English speaking
* Scheduled for induction of labor at the George Washington University Hospital

Exclusion Criteria:

* < 18 years of age
* Does not speak English
* Not scheduled for an induction of labor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Knowledge of Induction of Labor | 3 minute knowledge based questionnaire given to both arms prior to meeting with a provider (midwife or obstetrician).
  Evaluating if a 3-minute educational video changes patients' baseline knowledge of the induction of labor process when compared to patients' who receive traditional care via a questionnaire.

SECONDARY OUTCOMES:
Satisfaction with Induction of Labor Process | 3 minute satisfaction questionnaire given to both arms 24 to 48 hours after delivery at a time convenient for them.
  Evaluating if a 3-minute educational video changes patients' overall satisfaction with their delivery course when compared to patients' who received the standard care via a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sara H Rahman, MD, Study Director — Dr.
Locations (1):
- George Washington University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rahman S, Kripalani S, Keegan E, Sparks A, Amdur R, Moawad G, Sheth S, Klebanoff J. An educational video's impact on the induction of labor experience: a randomized controlled trial. Am J Obstet Gynecol MFM. 2022 Jan;4(1):100495. doi: 10.1016/j.ajogmf.2021.100495. Epub 2021 Sep 24. PMID 34571210

DOCUMENTS (3):
  • Informed Consent Form (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT04537260/ICF_000.pdf
  • Study Protocol (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT04537260/Prot_001.pdf
  • Statistical Analysis Plan (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT04537260/SAP_002.pdf